CLINICAL TRIAL: NCT06974981
Title: Leveraging Lung Cancer Screening to Optimize Screening Outcomes and COPD Management: COPD in LCS Registry
Acronym: COPD in LCS
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: iRISID-2024-1246
Record Dates: First submitted 2025-03-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: COPD - Chronic Obstructive Pulmonary Disease
Keywords: The COPD in LCS Registry will identify and characterize individuals who have functional or radiographic evidence of COPD and are receiving lung cancer screening
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The COPD in LCS Registry will identify and characterize individuals who have functional or radiographic evidence of COPD and are receiving lung cancer screening. Clinical information will be obtained from study participants including symptom burden, lung cancer risk, spirometry, imaging characteristics, and peripheral blood eosinophils.

ELIGIBILITY:
Inclusion Criteria:

* • * Eligible for lung cancer screening by USPSTF 2021 criteria including age 50-80 years and currently or formerly smoking with at last 20 pack-years of smoking history at the time of consent

  * Willingness to participate in an observational clinical trial and to be contacted about future ancillary studies that could include interventional clinical trials
  * Ability to tolerate study procedures
  * Ability to provide informed consent
  * Clinical Lung Cancer Screening CT performed at the University of Michigan within the last year
  * Meets one of the three following criteria: 1) Prior Diagnosis of COPD in the EMR 2) Prior pulmonary function meeting criteria for COPD (FEV1/FVC ≤ 0.70) or 3) LAA>1% on lung cancer screening CT scan

Exclusion Criteria:

* The presence of a respiratory condition other than COPD or asthma, or of a comorbid condition that in the judgment of the investigator may be the principal cause of respiratory symptoms (e.g. dyspnea or decreased exercise tolerance)Severe asthma, which is defined as any of the following:

  * Current (i.e. at the time of the visit) GINA Step 4 or higher therapy (medium dose ICS/LABA or high dose ICS or add-on LAMA; medium dose = >250 fluticasone propionate =100 fluticasone furoate, >200 beclomethasone, >400 budesonide, >220 mometasone). We will accept low-dose ICS/LABA or medium dose ICS or
  * 3 or more unscheduled healthcare visits (provider/urgent care/ER) for asthma in the past 12 months or
  * One asthma hospitalization in the past 12 months

    * Concurrent participation in a therapeutic trial where treatment is blinded
    * Active pregnancy. Documentation of birth control will be required for pre-menopausal women
    * Cognitive dysfunction that prevents the participant from completing study procedures
    * BMI > 35 kg/m2 at baseline, due to the effects of body weight on CT scan quality
    * Current illicit substance abuse, including cannabis smoking
    * Any illness expected to cause mortality in the next 3 years
    * Any implanted metallic devices or prosthesis above the waist that could degrade thoracic CT scan quality
    * History of thoracic radiation or thoracic surgery with resection of lung tissue
    * Participants who present with an acute exacerbation of COPD, either solely participant-identified or that has been clinically treated, in the last 30 days can be rescreened for the study once the 30-day window from end of drug therapy has passed
    * Participants who present with current use of acute antibiotics or steroids can be rescreened for the study >= 30 days after discontinuing acute antibiotics/steroids. This restriction does not apply to participants who are on chronic prednisone therapy of <10 mg per day or <20 mg every other day or participants who are currently on chronic, prophylactic, or suppressive antibiotic therapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for lung cancer screening due to their age and history of tobacco use, and have COPD, chronic bronchitis, or emphysema
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
COPD diagnosis based on meeting spirometric criteria | 2 years
  Will be based on meeting spirometric criteria for COPD (FEV^1/FVC =< 0.7) and have >1% low attenuation area on low-dose CT for LCS
Accrual rate | 2 years
  Will be reported using percentages and 95% exact confidence intervals.
Intervention compliance rate | 2 years
  Will be reported using percentages and 95% exact confidence intervals.
Follow-up retention rate | 2 years
  Will be reported using percentages and 95% exact confidence intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Racial Differences in Lung Cancer Screening Beliefs and Screening Adherence. Clinical lung cancer. 2021;22(6):570-8. doi: — https://doi.org/10.1016/j.cllc.2021.06.003
- See also: Nonmalignant Surgical Resection Among Individuals with Screening-Detected Versus Incidental Lung Nodules. Clinical lung cancer. 2023. doi: — https://doi.org/10.1016/j.cllc.2023.12.006